CLINICAL TRIAL: NCT00311181
Title: Phase 4 Study That Compares the DFT (Defibrillation Threshold) Efficacy of 3 Different Membrane Time Constant Based Biphasic Defibrillation Waveforms
Brief Title: POWER (Pulse Width Optimized Waveform Evaluation Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CRD 324
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Sudden Cardiac Death
Keywords: ICD; Defibrillation; ULV; Tuned
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Defibrillators, Implantable; Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2.5/3.5/4.5 ms defibrillation waveform (Experimental)
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT-D)

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT-D) — Patients that are indicated for an ICD or CRT-D receive one of these devices.

SUMMARY:
The objective of this study is to compare the ULV (Upper Limit of Vulnerability)/DFT (Defibrillation Threshold) efficacy between the 2.5, 3.5 and 4.5 ms membrane time constant based biphasic defibrillation waveforms. This comparison will result in identifying the optimal membrane time constant when programming the "tuned" defibrillation waveform.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) continues to be a significant cause of cardiac mortality with annual deaths ranging from 250,000 to 400,000 in the United States. Accordingly, implantable cardioverter-defibrillators (ICD's) have proven to be an important therapeutic option for patients susceptible to SCD. Successful therapy and generator longevity are greatly dependent on proper defibrillation threshold (DFT) determination.

All modern ICD's utilize a biphasic waveform for defibrillation. It has been clearly shown that biphasic waveforms reduce the energy required for internal defibrillation of the heart. However, there is no consensus on which pulse widths are best for defibrillation.

St. Jude Medical ICD's (implantable cardioverter defibrillators) have programmable pulse widths, which allow the physician multiple options in dealing with ICD patients. By implanting ICD's with programmable pulse widths, this study utilizes the Tissue RC Resistance/Capacitance) model to try to identify the optimal pulse widths.

To determine the efficacy of an optimal membrane time constant estimate for the "tuned" waveform, defibrillation testing must be performed. Upper limit of vulnerability (ULV) has been proposed as an alternative means of predicting the DFT and it has been shown that ULV guided DFT testing can achieve a defibrillation success rate of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for ICD/CRT-D implantation.
* Patient has a compatible transvenous defibrillation lead system.
* Patient has had an echocardiogram, MUGA, or cath procedure within 6 months of ICD/CRT-D implant.
* Patient is able to tolerate ULV guided DFT testing.

Exclusion Criteria:

* Patient has a mechanical valve in the tricuspid position.
* Patient has epicardial defibrillation electrodes.
* Patient is pregnant.
* Patient is less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shephal Doshi, MD, Principal Investigator — Pacific Heart Institute
Locations (2):
- United States (2):
  - Baptist Medical Center Montclair, Birmingham, Alabama
  - Pacific Heart Institute, Santa Monica, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 217
Completed | 121
Not Completed | 96
Not completed — Final DFTs were not obtained | 96

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 160
Region of Enrollment [Number; unit: participants]
  United States | 217

OUTCOME MEASURES:

1. Primary Outcome: Defibrillation Thresholds (DFTs) (3.5 ms Waveform)
Time Frame: Implant
Measure: Mean (Standard Error); unit: Volts
Arm/Group | Group 1
Number analyzed (Participants) | 121
Volts | 427 (11)

2. Primary Outcome: DFT (2.5 ms Waveform)
Time Frame: Implant
Measure: Mean (Standard Error); unit: Volts
Arm/Group | Group 1
Number analyzed (Participants) | 121
Volts | 454 (11)

3. Primary Outcome: DFT (4.5 ms Waveform)
Time Frame: Implant
Measure: Mean (Standard Error); unit: Volts
Arm/Group | Group 1
Number analyzed (Participants) | 121
Volts | 435 (11)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/217
Other Adverse Events (participants affected / at risk) | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No